CLINICAL TRIAL: NCT03545854
Title: Determination of Relationship Between Volume and Dispersion of Local Anesthetic on Ultrasound-guided Erector Spinae Plane Block in Cadavers
Brief Title: Dispersion of Local Anesthetic on the Erector Spinae Plane Block in Cadavers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Vaz Perez, Medical Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Erector Spinae Plane Block
Record Dates: First submitted 2018-05-12; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Nerve Block

STUDY DESIGN:
Intervention Model Description: The cadavers will be randomized to receive the intervention (Erector Spinae Plane Block) on different levels (Vertebral level - T3, T12 and L4) and different volumes (10, 20 and 30ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- T3 10ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 10ml of coloring solution at the T3 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- T3 20ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 20ml of coloring solution at the T3 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- T3 30ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 30ml of coloring solution at the T3 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- T12 10ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 10ml of coloring solution at the T12 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- T12 20ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 20ml of coloring solution at the T12 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- T12 30ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 30ml of coloring solution at the T12 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- L4 10ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 10ml of coloring solution at the L4 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- L4 20ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 20ml of coloring solution at the L4 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- L4 30ml (Experimental): The cadaver will receive an ultrasound-guided Erector Spinae Plane Block with 30ml of coloring solution at the L4 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Ultrasound guided injection of coloring solution (methylene blue diluted in water) with a 18G echogenic tuohy needle deep to the plane of the erector spinae muscles.

SUMMARY:
This study aims to better understand the dispersion of local anesthetic on the Erector Spinae Block, a new technique developed for analgesia. It consists on injection of local anesthetic around the posterior muscles of the Spine. In this study, the investigators will make the injection with coloring solution on cadavers and by dissection will note the dispersion of the solution according to injectate volume. The investigators hypothesize more volume allows bigger spread and will allow new indications of this technique in perioperative analgesia and treatment of chronic Pain

DETAILED DESCRIPTION:
The study's methodology will include performing ultrasound guided erector spinae block in cadavers included in the study according to eligibility criteria. After signing of written consent form, the participants will be randomized on the height of the block (vertebral level - T3, T12 and L4) and the volume to be injected (10, 20 and 30ml). The block will be performed by experienced physicians on the technique by ultrasound guidance and fixed pressure measured with an in-line pressure monitor (15 psi) with the cadaver in the lateral position. The cadavers will be submitted to autopsy by standard thoracoabdominal midline incision, with the viscera removed for analysis. The cadavers will have their paraspinal muscles removed (quadratus lumborum and psoas major), the medial parietal pleura opened and the number of levels with colored solution registered, noting the spread to ventral rami of spinal nerves and to the paravertebral space.

ELIGIBILITY:
Inclusion Criteria:

* Fresh Cadavers (not subject to formaldehyde fixation process or frozen > 24h)
* Age > 18 years
* Written informed consent signed by responsible party
* Height > 150cm and < 190cm

Exclusion Criteria:

* Previous spinal surgery
* Severe spinal deformity
* BMI > 35 kg/m2
* Absence of a responsible party to sign the written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Spread of Coloring Solution secondary to volume injected and vertebral level of injection | 3 hours
  Observation of coloring solution around the spinal nerves as they exit the vertebral foramen. Comparison of number of spinal nerves colored according to the volume injected and injection site.

SECONDARY OUTCOMES:
Spread of coloring solution to paravertebral space | 3 hours
  Observation of coloring solution on the paravertebral space. Comparison of number of levels of the paravertebral space colored according to volume injected and injection site.

CONTACTS AND LOCATIONS:
Overall Officials: Andre L Casale, MD, Principal Investigator — Post Graduate
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The research results will be published on indexed scientific journals, maintaining participant identity confidential

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Elsharkawy H, Pawa A, Mariano ER. Interfascial Plane Blocks: Back to Basics. Reg Anesth Pain Med. 2018 May;43(4):341-346. doi: 10.1097/AAP.0000000000000750. PMID 29561295
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Leyva FM, Mendiola WE, Bonilla AJ, Cubillos J, Moreno DA, Chin KJ. Continuous Erector Spinae Plane (ESP) Block for Postoperative Analgesia after Minimally Invasive Mitral Valve Surgery. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2271-2274. doi: 10.1053/j.jvca.2017.12.020. Epub 2017 Dec 12. No abstract available. PMID 29336964
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Gaio-Lima C, Costa CC, Moreira JB, Lemos TS, Trindade HL. Continuous erector spinae plane block for analgesia in pediatric thoracic surgery: A case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):287-290. doi: 10.1016/j.redar.2017.11.010. Epub 2018 Jan 19. English, Spanish. PMID 29370900
- [Background] Nandhakumar A, Nair A, Bharath VK, Kalingarayar S, Ramaswamy BP, Dhatchinamoorthi D. Erector spinae plane block may aid weaning from mechanical ventilation in patients with multiple rib fractures: Case report of two cases. Indian J Anaesth. 2018 Feb;62(2):139-141. doi: 10.4103/ija.IJA_599_17. PMID 29491521
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771
- [Background] Aksu C, Gurkan Y. Ultrasound-guided bilateral erector spinae plane block could provide effective postoperative analgesia in laparoscopic cholecystectomy in paediatric patients. Anaesth Crit Care Pain Med. 2019 Feb;38(1):87-88. doi: 10.1016/j.accpm.2018.03.008. Epub 2018 Apr 6. No abstract available. PMID 29630940
- [Background] Restrepo-Garces CE, Chin KJ, Suarez P, Diaz A. Bilateral Continuous Erector Spinae Plane Block Contributes to Effective Postoperative Analgesia After Major Open Abdominal Surgery: A Case Report. A A Case Rep. 2017 Dec 1;9(11):319-321. doi: 10.1213/XAA.0000000000000605. PMID 28727597
- [Background] Tulgar S, Senturk O. Ultrasound guided low thoracic erector spinae plane block for postoperative analgesia in radical retropubic prostatectomy, a new indication. J Clin Anesth. 2018 Jun;47:4. doi: 10.1016/j.jclinane.2018.02.013. Epub 2018 Mar 5. No abstract available. PMID 29518667
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Ueshima H, Hiroshi O. RETRACTED: Transapical transcatheter aortic valve implantation performed with an erector spinae plane block. J Clin Anesth. 2018 May;46:84. doi: 10.1016/j.jclinane.2018.02.001. Epub 2018 Feb 3. No abstract available. PMID 29414628 (Retraction: PMID 35537956 J Clin Anesth. 2022 Sep;80:110801)
- [Background] Ueshima H. RETRACTED: Pneumothorax after the erector spinae plane block. J Clin Anesth. 2018 Aug;48:12. doi: 10.1016/j.jclinane.2018.04.009. Epub 2018 Apr 21. No abstract available. PMID 29684727 (Retraction: PMID 35393181 J Clin Anesth. 2022 Aug;79:110763)
- [Background] Ueshima H, Hiroshi O. RETRACTED: Spread of local anesthetic solution in the erector spinae plane block. J Clin Anesth. 2018 Mar;45:23. doi: 10.1016/j.jclinane.2017.12.007. Epub 2017 Dec 16. No abstract available. PMID 29258057 (Retraction: PMID 35551829 J Clin Anesth. 2022 Sep;80:110834)
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152